CLINICAL TRIAL: NCT06611059
Title: Design of Patient Specific Guides (PSG) for Reverse Shoulder Arthroplasty
Acronym: PSG
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-PSG-2023-107; IIBSP-PSG-2023-107 (Registry Identifier: Clinical Research Ethics Committee)
Record Dates: First submitted 2023-12-19; First posted 2024-09-24 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Proximal Humeral Fracture
Keywords: reverse shoulder arthroplasty; patient specific guide; 3D
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- in-hospital designed patient specific guide
  Interventions: Device: PSG

INTERVENTIONS:
Device: PSG — Two replicas of each scapula are made. The scapulae are drilled with a commercial guide and with an in-house guide separately
  Other Names: Patient Specific Guides

SUMMARY:
This is a two steps observational study

In the first part we will compare the accuracy of the commercial guide against a in-hospital designed patient specific guide. As a secondary goal, the problems detected during the design phase will be described.

Once the accuracy of the guide is acceptable, we will implant the glenosphere of future patients using the PSG guide following the same engineering design process.

DETAILED DESCRIPTION:
Reverse shoulder arthroplasty is a treatment for both non-synthesizable fractures and arthropathy degenerative. This implant is based on two main components: glenosphere and stem. The stem in turn is integrated in its upper part by a polyethylene that reduces the friction torque between the glenosphere and the stem.

Correct positioning of the glenosphere is critical for functionality and survival of the implant. Malpositioning of glenosphere can be related to:

In recent years, given the

* The scapula is a flat bone, without any reference axis;
* Surgical approaches expose only the glenoid cavity, with few bone landmarks;
* The humerus and deltoid make access to the glenoid difficult;
* The morphology of the scapula is very variable.

Preoperative planning even without PSG improves the positioning accuracy of the guide in the glenoid. In glenoids with only a slight deformity, PSGs improve the accuracy of the guide entry point (&lt;1 mm error, compared to &gt; 4 mm under visual control) and orientation (&lt; 3◦ error compared to &gt; 7◦). In glenoids with more significant deformities, planning also showed superiority.

ELIGIBILITY:
Inclusion Criteria:

* Patient with proximal humerus fracture candidate for reversed shoulder arthroplasty
* Patient with degenerative arthropathy candidate for reversed shoulder arthroplasty

Exclusion Criteria:

* Previous surgeries on the proximal humerus or glenoid
* No desire to participate in the study
* Lack of ability to accept the study (tutored patients)
* Open fractures

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * Patient with proximal humerus fracture candidate for reversed shoulder arthroplasty
  * Patient with degenerative arthropathy candidate for reversed shoulder arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-01-23 (Actual)

PRIMARY OUTCOMES:
Difference in glenoid center | months
  Difference in glenoid center (mm): distance between the points of entry on the surface of the scapula, the planned center versus the finally drawn
Glenoid version deviation (α) | months
  Glenoid version deviation (α): defined as the angle between the real trajectory of the drilling and the scapular anatomical plane, projected about the axis of neutral inclination (defined as that which goes from the center of the glenoid to the trigonum spinae).
Glenoid inclination deviation (β) | months
  Glenoid inclination deviation (β): defined as the angle between the actual milling path and the plane of the neutral tilt axis, projected on the SP axis

CONTACTS AND LOCATIONS:
Overall Officials: A. Millan, Principal Investigator — Orthopedic and Trauma Dept. / Trauma Unit; A. Toro, Study Director — Orthopedic and Trauma Dept. / Trauma Unit
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Gauci MO. Patient-specific guides in orthopedic surgery. Orthop Traumatol Surg Res. 2022 Feb;108(1S):103154. doi: 10.1016/j.otsr.2021.103154. Epub 2021 Nov 24. PMID 34838754
- [Background] Gonzalez JF, Alami GB, Baque F, Walch G, Boileau P. Complications of unconstrained shoulder prostheses. J Shoulder Elbow Surg. 2011 Jun;20(4):666-82. doi: 10.1016/j.jse.2010.11.017. Epub 2011 Mar 21. No abstract available. PMID 21419661
- [Background] Jacquot A, Gauci MO, Chaoui J, Baba M, Deransart P, Boileau P, Mole D, Walch G. Proper benefit of a three dimensional pre-operative planning software for glenoid component positioning in total shoulder arthroplasty. Int Orthop. 2018 Dec;42(12):2897-2906. doi: 10.1007/s00264-018-4037-1. Epub 2018 Jul 2. PMID 29968136
- [Background] Berhouet J, Gulotta LV, Dines DM, Craig E, Warren RF, Choi D, Chen X, Kontaxis A. Preoperative planning for accurate glenoid component positioning in reverse shoulder arthroplasty. Orthop Traumatol Surg Res. 2017 May;103(3):407-413. doi: 10.1016/j.otsr.2016.12.019. Epub 2017 Feb 24. PMID 28238965
- [Background] Gauci MO, Boileau P, Baba M, Chaoui J, Walch G. Patient-specific glenoid guides provide accuracy and reproducibility in total shoulder arthroplasty. Bone Joint J. 2016 Aug;98-B(8):1080-5. doi: 10.1302/0301-620X.98B8.37257. PMID 27482021
- [Background] Iannotti JP, Walker K, Rodriguez E, Patterson TE, Jun BJ, Ricchetti ET. Accuracy of 3-Dimensional Planning, Implant Templating, and Patient-Specific Instrumentation in Anatomic Total Shoulder Arthroplasty. J Bone Joint Surg Am. 2019 Mar 6;101(5):446-457. doi: 10.2106/JBJS.17.01614. PMID 30845039
- [Background] Levy JC, Everding NG, Frankle MA, Keppler LJ. Accuracy of patient-specific guided glenoid baseplate positioning for reverse shoulder arthroplasty. J Shoulder Elbow Surg. 2014 Oct;23(10):1563-7. doi: 10.1016/j.jse.2014.01.051. Epub 2014 Apr 13. PMID 24739791
- [Background] Cabarcas BC, Cvetanovich GL, Espinoza-Orias AA, Inoue N, Gowd AK, Bernardoni E, Verma NN. Novel 3-dimensionally printed patient-specific guide improves accuracy compared with standard total shoulder arthroplasty guide: a cadaveric study. JSES Open Access. 2019 Jun 15;3(2):83-92. doi: 10.1016/j.jses.2019.04.001. eCollection 2019 Jul. PMID 31334434
- [Background] Dallalana RJ, McMahon RA, East B, Geraghty L. Accuracy of patient-specific instrumentation in anatomic and reverse total shoulder arthroplasty. Int J Shoulder Surg. 2016 Apr-Jun;10(2):59-66. doi: 10.4103/0973-6042.180717. PMID 27186057
- [Background] Cabarcas BC, Cvetanovich GL, Gowd AK, Liu JN, Manderle BJ, Verma NN. Accuracy of patient-specific instrumentation in shoulder arthroplasty: a systematic review and meta-analysis. JSES Open Access. 2019 Sep 18;3(3):117-129. doi: 10.1016/j.jses.2019.07.002. eCollection 2019 Oct. PMID 31709351
- [Background] Villatte G, Muller AS, Pereira B, Mulliez A, Reilly P, Emery R. Use of Patient-Specific Instrumentation (PSI) for glenoid component positioning in shoulder arthroplasty. A systematic review and meta-analysis. PLoS One. 2018 Aug 22;13(8):e0201759. doi: 10.1371/journal.pone.0201759. eCollection 2018. PMID 30133482